CLINICAL TRIAL: NCT00999154
Title: Diet-Induced-Obesity Resistant Phenotypes in Humans
Status: Terminated | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090238; 09-DK-0238
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2012-10-22

CONDITIONS: Healthy Volunteers
Keywords: Energy Expenditure; Dietary Intake; Physical Activity; Body Weight Regulation; Sedentary; HV; Healthy Volunteer
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Obesity is the result of many factors, including genetics and lifestyle, such as over-eating high-calorie foods and not being physically active. Obesity affects approximately one third of adults in the United States. Researchers often study individuals who are already overweight and obese, but another approach is to examine people who stay thin despite eating whatever they want and not exercising. Studying these thin individuals will enhance understanding of why some people become obese and others do not, which may lead to novel treatments for obesity.

Objective:

- To study the metabolism, body composition, body temperature, physical activity, and blood chemistries of healthy lean adults before and after adding 1,000 extra Calories per day to their normal diet.

Eligibility:

- Healthy adults, 30 to 50 years of age, who have never been overweight after adolescence, who are currently weight-stable, sedentary, and eating without restrictions.

Design:

- The entire study will take about 9 weeks and will include the following outpatient and inpatient visits:

<TAB>- Outpatient screening visit and monitoring: Physical examination and blood test at screening; then, one week of physical activity monitoring (e.g., with a pedometer-like device called an accelerometer) and completing a food diary.

<TAB>- Baseline inpatient visit (5 days): Volunteers will eat a normal diet to maintain body weight. Energy expenditure, body composition, physical fitness, activity level, and eating behavior will be measured. Urine and blood samples will be taken. Volunteers may go home for the weekend or stay at the metabolic clinical research unit (MCRU).

<TAB>- Inpatient feeding week 1 (5 days): Volunteers will eat a normal diet plus milkshakes for added calories. All the same measurements during the baseline week visit will be repeated.

<TAB>- Outpatient feeding weeks 2 3: Volunteers will eat breakfast at the MCRU everyday for the next 2 weeks and take prepared meals home with them (volunteers may also stay at the MCRU for the 2 weeks if they prefer). Volunteers will drink a non-radioactive (heavy) water called doubly labeled water to measure energy expenditure in their normal living environment Daily urine samples will be collected.

<TAB>- Inpatient feeding week 4 (5 days): Volunteers will continue eating a normal diet plus milkshakes for added calories. This stay and measurement is identical to inpatient feeding week 1.

- Volunteers will be contacted at 6 and 12 months to assess any changes in body weight, diet, and physical activity.

DETAILED DESCRIPTION:
While many obesity studies focus on the individuals who are already overweight and obese, a complementary approach to understand such a common disease is to define the mechanisms which allow some lean individuals to resist weight gain. The predominant cause of human obesity is the inheritance of genes favoring fat storage and efficient energy utilization interacting with an obesogenic environment, characterized by readily available, energy-dense food and sedentary lifestyle. However, a persistent percentage (about 30%) of the US adult population remains thin (BMI <23 kg/M(2)). While some of these individuals maintain their weight by vigilantly controlling their diet, exercising or taking medication(s), others may have the ability to remain thin despite an excessive energy intake and without volitional exercise. To identify these individuals and define their phenotypes will provide unique insights into energy and body weight homeostasis, and may yield novel approaches for treating obesity.

In this natural history protocol, we will recruit and characterize a cohort of constitutionally lean and healthy adult volunteers (age 25-50, BMI 18.5-25 kg/M(2)) who do not have pathological or exogenous factors that are known to stimulate energy expenditure, suppress food intake, or decrease absorption. We will recruit volunteers who are weight-stable, sedentary, and non-restrictive eaters, characterize their free-living dietary and physical activity energy expenditure using food records and portable accelerometers, respectively. Using an inpatient controlled setting, we will carefully characterize the details of their 24-hr energy metabolism, body composition, core and skin temperatures, and blood chemistries while they are on a one-week metabolic diet adjusted to maintain his/her body weight (baseline) vs. another week of higher energy intake level (1000 extra kcal per day above their baseline). Overfeeding will continue for two more weeks in the outpatient setting with all meals provided by our metabolic kitchen, followed by the fourth week of overfeeding and repeated measurements back in the inpatient setting. We hypothesize that spontaneous changes in energy expenditure and/or calorie intake may differ between individuals, and such difference may explain the ability for some to resist body gain. The accruals of humans with obesity-resistant phenotypes will significantly enhance our understanding of the mechanisms of energy homeostasis and identify potential novel regulators for controlling obesity.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Healthy normal men and women between 25-50 years of age;
  2. BMI between 18.5 and 25.0 kg/M(2);
  3. Self-reported as having had trouble gaining weight, who doing little or no exercise, self-described or by friends or family members as an overeater, and who have never tried to lose weight.

EXCLUSION CRITERIA:

1. A self-reported history of overweight after the age of 18, other than during pregnancy for women;
2. Recent weight changes >2% of current body weight in the last 6 months;
3. Current or past history of eating disorders such as binge eating, anorexia nervosa, or bulimia, by psychological evaluations;
4. Current or past history of intentional weight loss by self-report, other than postpartum weight loss;
5. High physically demanding occupations or volitional exercise >20 total minutes/day of moderate intensity or higher (as measured by sweating), >2 days/week, by self-report;
6. Significant dietary limitations (multiple food allergies/intolerances, vegan diet, etc.) that may affect absorption and body weight, or special dietary requirements that are difficult to accommodate with by study diets;
7. Significant physical limitations that may preclude completing the majority of the tests in this study;
8. Current pregnancy, recent pregnancy (<3 years), current/recent breast feeding (<1 year), or perimenopausal status. During the study, women may be asked to use birth control and will undergo repeated pregnancy testing. Subjects who refuse these tests will be excluded;
9. Current or past medical conditions that are known to affect energy metabolism and body weight regulations, including HIV/AIDS, cancer, cardiac ischemia, dyslipidemia, thyroid and parathyroid disorders, hypo- or hypertension, diabetes (type 1 or type 2) or impaired glucose tolerance, congenital or acquired lipodystrophy, hepatic, renal, neuromuscular, celiac disease and other malabsorptive conditions, known genetic disorders that alter lipid metabolism, or cardiac failure as assessed by history and physical exam;
10. Any psychiatric condition (including psychosis) or personality disorder as judged by the PI or Co-PI that would impede participation in the study;
11. Smoking (currently or within the past year), excessive caffeine (>500 mg/day) and/or alcohol intake (>2 drinks/day for men, > 1 drink/day for women), as assessed by self reports and serum thiocyanate;
12. Taking narcotics, cocaine, or marijuana which would alter metabolism (positive urine toxicology screen)
13. Any use of medications or nutritional supplements known to increase EE, depress food intake, or affect absorption;
14. Unwilling or unable to give informed consent;
15. Any other clinical or sub-clinical conditions not mentioned above that are considered by the investigators as significant exclusions for the study.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2009-09-19; Study Completion 2012-10-22

CONTACTS AND LOCATIONS:
Overall Officials: Kong Y Chen, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Comuzzie AG, Allison DB. The search for human obesity genes. Science. 1998 May 29;280(5368):1374-7. doi: 10.1126/science.280.5368.1374. PMID 9603720
- [Background] Coleman DL. Obesity genes: beneficial effects in heterozygous mice. Science. 1979 Feb 16;203(4381):663-5. doi: 10.1126/science.760211.